CLINICAL TRIAL: NCT03179722
Title: Studying the Impact of a Medication Use Evaluation by the Community Pharmacist
Acronym: SIMENON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joke Wuyts (Other)
Collaborators: Association of Belgian Pharmacies (APB) (Unknown)
Responsible Party: Sponsor-Investigator, Joke Wuyts, PharmD, KU Leuven
Organization: KU Leuven (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SIMENONv3
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Aging
Keywords: Aging; Drug-related problems; Medication review; Community pharmacist; Medication use
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Parallel group intervention study. In a subset of 140 patients, a pre-post study design is used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Frenchspeaking patients (Experimental): Intervention: Medication review
  Interventions: Behavioral: Medication review
- Intervention group: Dutchspeaking patients (Experimental): Intervention: Medication review Intervention: Dutchspeaking patients are also invited to participate to Additional data collection: questionnaires
  Interventions: Behavioral: Medication review; Behavioral: Additional data collection: questionnaires

INTERVENTIONS:
Behavioral: Medication review — The intervention consists of a medicines use review provided by community pharmacists in Belgium. A medicines use review is a medication review type 2a in which both a patient interview and dispensing data are used as information sources to identify drug-related problems with a specific focus on the medicines use of the patient.
  Other Names: Medication use review; Medication review type 2a; Intermediate medication review
Behavioral: Additional data collection: questionnaires — Pre-post study design.
  At three timepoints, data is collected:
  * before the medication review (T-1week)
  * during the review (Tweek 3)
  * after the review (Tweek12) The questionnaire provide data for the outcomes: medication related quality of life, adherence questionnaire, service satisfaction, use of emergency health services, self-management
  Arms: Intervention group: Dutchspeaking patients

SUMMARY:
In this intervention study, 75 Belgian community pharmacies each recruit 12 patients for an intermediate medication review. For each patient, the identified drug-related problems and subsequent interventions are registered using the PharmDisc classification. In a subset of Dutch speaking patients, a pretest-posttest single group design is used to measure the impact of this review on patient related outcomes using questionnaires. The primary outcome is the medication related quality of life, measured via the living with medicines questionnaire. Other patient reported outcomes include adherence, self-management, patient satisfaction, fall incidents and use of emergency healthcare services. Medication records are also collected to objectively measure adherence before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 70 years or older
* Use five or more drugs on a regular basis (prescription or non-prescription drugs)
* Live in the ambulatory setting
* Obtain his medication from this pharmacy on a regular basis

Exclusion Criteria:

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 453 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2017-10-11 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Drug-related problems & interventions | One timeframe: during the medication review
  Using the validated PharmDisc classification tool
Change in medication related quality of life | Three timepoints: Before the review, during review (week 3), after the review (week 12)
  using the Living with medicines questionnaire

SECONDARY OUTCOMES:
Change in adherence | 9 months before and after the intervention
  using dispensing data
Change in adherence | Two timepoints: Before the review, after the review (week 12)
  using the PROMAS questionnaire
Change in self-management | Two timepoints: Before the review, after the review (week 12)
  using the PAM questionnaire
Change in use of emergency healthcare services & fall incidents | Two timepoints: Before the review, after the review (week 12)
  using own questions
Satisfaction with the new service | One timepoint: during the review (week 3)
  Using the PSPSQ2 questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wuyts J, Maesschalck J, De Wulf I, Foubert K, Boussery K, De Lepeleire J, Foulon V. Studying the impact of a medication use evaluation for polymedicated older patients by the community pharmacist (SIMENON): study protocol. BMC Health Serv Res. 2018 Aug 8;18(1):623. doi: 10.1186/s12913-018-3440-z. PMID 30089523
- See also: Protocol Abstract for the PCNE conference 2017 (DOI: 10.1007/s11096-017-0462-2) — https://link.springer.com/article/10.1007/s11096-017-0462-2